CLINICAL TRIAL: NCT07292220
Title: Investigation of Neurofilament Light Chain (NfL) Levels in Newborns Diagnosed With Hypoxic Ischemic Encephalopathy: A Case-Control Study
Brief Title: A Study of a Blood Marker in Newborns With Brain Injury Caused by Lack of Oxygen at Birth
Status: Not yet recruiting | Type: Observational
Sponsor: Mustafa Gürkan (Other)
Responsible Party: Sponsor-Investigator, Mustafa Gürkan, assistant doctor, Kırıkkale University
Organization: Kırıkkale University (Other)
Other Study IDs: kırıkkale medical university
Record Dates: First submitted 2025-11-13; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Hypoxic-ischemic encephalopathy (HIE); Neurofilament light chain (NfL); Newborn; Therapeutic hypothermia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — In this study, only venous blood samples collected intravenously from participants will be used. The serum fraction obtained from the blood samples will be analyzed to measure neurofilament light chain (NfL) levels. No genetic analysis will be performed as part of this study, and no DNA, RNA, or cellular material isolation is planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- case: control case

SUMMARY:
Perinatal asphyxia is a significant health problem with an incidence of 1 to 8 per 1,000 live births and can lead to serious morbidity and mortality during the neonatal period. One of its most severe consequences is hypoxic-ischemic encephalopathy (HIE), a condition that causes irreversible damage to the newborn brain due to hypoxia and ischemia. HIE is one of the leading causes of long-term neurological sequelae. Therapeutic hypothermia initiated within the first six hours after birth has been shown to significantly reduce both mortality and neurodevelopmental impairments associated with HIE. However, biomarkers that can reliably predict individual treatment response or objectively demonstrate the severity of brain injury at an early stage remain limited.

Neurofilament light chain (NfL) is a protein found within the cytoskeletal structure of myelinated axons. When axonal injury occurs, NfL is released into the interstitial space and subsequently enters the cerebrospinal fluid and systemic circulation, where it can be measured. Increased NfL levels have been identified in a variety of neurological conditions, including neurodegenerative disorders and traumatic brain injury. Recent findings show that both cerebrospinal fluid and serum/plasma NfL levels are elevated in newborns diagnosed with HIE, supporting its potential role as a biochemical marker of axonal injury.

The primary aim of this study is to investigate the time-dependent changes in serum NfL levels in newborns diagnosed with HIE and undergoing therapeutic hypothermia, and to evaluate the relationship between these changes, clinical findings, and neuroimaging results. For this purpose, serum NfL levels were measured at four specific time points: within the first six hours after birth (preferably cord blood), upon reaching the target cooling temperature (approximately 12-24 hours), during the rewarming phase (72-96 hours), and on the day of magnetic resonance imaging (preferably day seven). The results are expected to provide insights into the prognostic utility of NfL in HIE and contribute to determining the optimal timing for clinical sampling.

The secondary objective of the study is to compare NfL levels of newborns diagnosed with HIE to those of a control group without HIE, thereby identifying potential cut-off values that may help distinguish between affected and unaffected infants.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a critical clinical condition arising from perinatal asphyxia, leading to acute-phase mortality and significant long-term neurological morbidity during the neonatal period. In recent years, therapeutic hypothermia has become the standard treatment approach for HIE, with proven effectiveness in reducing both mortality and severe neurodevelopmental sequelae. However, its therapeutic benefit is not consistent across all cases, and some newborns may still develop permanent neurological damage and developmental impairments despite receiving treatment. This highlights the need for reliable biomarkers that can reveal the extent of central nervous system injury in the early period, predict prognosis, and objectively assess treatment response.

Neurofilament light chain (NfL), a myelinated axon-specific structural protein released into the bloodstream following central nervous system injury, has gained increasing attention as a potential biomarker. Neurofilaments are abundant within axons and play a crucial role in radial growth during development, maintenance of axon caliber, and electrical signal conduction. They are intermediate filaments with a diameter of approximately 10 nm and are composed of four major subunits within the central nervous system: heavy, medium, and light neurofilament polypeptides, along with α-internexin.

In various pathological conditions, neurofilaments may accumulate in large quantities within neuronal cell bodies and proximal axons. Such accumulations are characteristic lesions in several neurological disorders, including motor neuron diseases, hereditary neuropathies, neurofilament inclusion disorders, giant axonal neuropathies, metabolic neuropathies, and degenerative motor neuron conditions. Although NfL levels are typically higher in cerebrospinal fluid than in blood, serum or plasma measurements are clinically advantageous due to their minimally invasive nature, reproducibility, and practical applicability. Accordingly, NfL has been widely investigated as a biomarker in both cerebrospinal fluid and blood for a range of neurodegenerative and neurological diseases.

In the neonatal population, clinical investigations have largely focused on HIE, where serum and plasma NfL levels have been associated with disease severity and long-term neurodevelopmental outcomes. Beyond HIE, NfL also shows potential prognostic value in preterm-related morbidities such as intraventricular hemorrhage, periventricular leukomalacia, and diffuse white matter injury. Moreover, its use is being explored as a biochemical indicator of perioperative neurological injury in infants undergoing cardiopulmonary bypass for congenital heart disease, as well as in neonatal sepsis and sepsis-associated encephalopathy.

Recent research has demonstrated significant associations between NfL levels and both magnetic resonance imaging findings and long-term neurodevelopmental outcomes in newborns with HIE treated with therapeutic hypothermia. These observations support the potential of NfL as a biomarker reflecting axonal injury and as a prognostic indicator. However, the number of studies that systematically compare NfL levels at different sampling time points remains limited, emphasizing the need to determine the optimal timing of measurement and to standardize its use in clinical practice.

The primary objective of this study is to measure NfL levels in blood samples obtained at defined time intervals after birth in order to assess the timing and extent of brain involvement. This will support early prognostic evaluation and contribute to the development of future diagnostic algorithms. The secondary objective is to compare infants diagnosed with HIE to a control group, thereby clarifying the extent of brain injury associated with HIE in the neonatal period.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns with a gestational age ≥36 weeks (term)
2. Diagnosis of hypoxic ischemic encephalopathy (HIE) based on clinical and/or laboratory findings
3. Diagnosis of stage I, stage II, or stage III HIE according to the Sarnat staging system
4. Therapeutic hypothermia (TH) treatment initiated within the first 6 hours after birth
5. Written consent obtained from the legal parent(s) for participation in the study

Exclusion Criteria:

1. Major congenital malformation or genetic syndrome (e.g., Trisomy 21, congenital heart disease)
2. Newborns with suspected sepsis, metabolic disease, or other systemic disease
3. Premature infants with a gestational age <36 weeks
4. Therapeutic hypothermia treatment not started on time or inadequately administered
5. Medical conditions preventing blood sampling (e.g., severe coagulopathy, circulatory instability)

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cases admitted to the Neonatal Intensive Care Unit of Kırıkkale University Faculty of Medicine Hospital with a diagnosis of hypoxic-ischemic encephalopathy (HIE) and started on therapeutic hypothermia (TH) treatment were prospectively recorded.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
1. Serum NfL Level at 0-6 Hours After Birth | Assessed at 0-6 hours after birth
  Measurement of serum neurofilament light chain concentration in blood collected within 0-6 hours after birth. Unit of Measure: pg/mL
Serum NfL Level at 12-24 Hours After Birth | Assessed at 12-24 hours after birth
  Measurement of serum NfL concentration in blood collected after achieving target therapeutic hypothermia temperature.Unit of Measure: pg/mL
Serum NfL Level at 72-96 Hours After Birth | Assessed at 72-96 hours after birth
  Measurement of serum NfL concentration during the rewarming phase.Unit of Measure: pg/mL
Serum NfL Level at Approximately Day 7 | Assessed at approximately 7 days after birth
  Measurement of serum NfL concentration on the day of clinically indicated brain MRI.Unit of Measure: pg/mL

SECONDARY OUTCOMES:
Sarnat Encephalopathy Stage at 0-6 Hours | Assessed at 0-6 hours after birth
  Clinical staging of hypoxic-ischemic encephalopathy severity using the standardized Sarnat scale.Unit of Measure: Stage I-III
Sarnat Encephalopathy Stage at 72-96 Hours | Time Frame: Assessed at 72-96 hours after birth
  Clinical staging of hypoxic-ischemic encephalopathy severity using the standardized Sarnat scale.Unit of Measure: Stage I-III
Sarnat Encephalopathy Stage at 12-24 Hours | Assessed at 12-24 hours after birth
  Clinical staging of hypoxic-ischemic encephalopathy severity using the standardized Sarnat scale.Unit of Measure: Stage I-III
Thompson Score at 0-6 Hours | Assessed at 0-6 hours after birth
  Neurological assessment using the standardized Thompson scoring system.Unit of Measure: Score (0-22)
Thompson Score at 12-24 Hours | Time Frame: Assessed at 12-24 hours after birth
  Neurological assessment using the standardized Thompson scoring system.Unit of Measure: Score (0-22)
Thompson Score at 72-96 Hours | Assessed at 72-96 hours after birth
  Neurological assessment using the standardized Thompson scoring system.Unit of Measure: Score (0-22)
Brain MRI Findings | Assessed at approximately 7 days after birth
  Evaluation of brain injury patterns based on routine MRI obtained during clinical care Unit of Measure: Qualitative classification (normal / abnormal)

CONTACTS AND LOCATIONS:
Locations (1):
- , Kirikkale University, Department of Pediatrics, Kirikkale, Kırıkkale, Yahşihan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: no end date

REFERENCES:
- [Background] Stull JW, Brown WH, Whiting FM. Some characteristics of metabolism of organochlorine compounds in the bovine. Fed Proc. 1973 Sep;32(9):1995-2002. No abstract available. PMID 4737695
- [Background] Shah DK, Ponnusamy V, Evanson J, Kapellou O, Ekitzidou G, Gupta N, Clarke P, Michael-Titus AT, Yip PK. Raised Plasma Neurofilament Light Protein Levels Are Associated with Abnormal MRI Outcomes in Newborns Undergoing Therapeutic Hypothermia. Front Neurol. 2018 Mar 5;9:86. doi: 10.3389/fneur.2018.00086. eCollection 2018. PMID 29556208
- [Background] Depoorter A, Neumann RP, Barro C, Fisch U, Weber P, Kuhle J, Wellmann S. Neurofilament Light Chain: Blood Biomarker of Neonatal Neuronal Injury. Front Neurol. 2018 Nov 20;9:984. doi: 10.3389/fneur.2018.00984. eCollection 2018. PMID 30524361
- [Background] Kyng KJ, Wellmann S, Lehnerer V, Hansen LH, Kuhle J, Henriksen TB. Neurofilament Light Chain serum levels after Hypoxia-Ischemia in a newborn piglet model. Front Pediatr. 2023 Jan 9;10:1068380. doi: 10.3389/fped.2022.1068380. eCollection 2022. PMID 36699314
- [Background] Rutherford M, Ramenghi LA, Edwards AD, Brocklehurst P, Halliday H, Levene M, Strohm B, Thoresen M, Whitelaw A, Azzopardi D. Assessment of brain tissue injury after moderate hypothermia in neonates with hypoxic-ischaemic encephalopathy: a nested substudy of a randomised controlled trial. Lancet Neurol. 2010 Jan;9(1):39-45. doi: 10.1016/S1474-4422(09)70295-9. Epub 2009 Nov 5. PMID 19896902
- [Background] Kurinczuk JJ, White-Koning M, Badawi N. Epidemiology of neonatal encephalopathy and hypoxic-ischaemic encephalopathy. Early Hum Dev. 2010 Jun;86(6):329-38. doi: 10.1016/j.earlhumdev.2010.05.010. Epub 2010 Jun 16. PMID 20554402